CLINICAL TRIAL: NCT06927336
Title: The Study on the Efficacy of tDCS Stimulation of the Cerebellum Combined With XingNaoJing Injection in Patients With Consciousness Disorders After Cranial Injury
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Liqing Yao, Department of rehabilitation medicine, the Second Affiliated Hospital of Kunming Medical University, The Second Affiliated Hospital of Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shen-PJ-Ke-2025-6
Record Dates: First submitted 2025-03-22; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: tDCS; Cerebellum; Brain Injury; Disturbance of Consciousness
MeSH Terms: conditions — Brain Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- tDCS combined with XingNaoJing treatment group (Experimental): The tDCS stimulation time was 20 minutes, once a day, 5 times a week, a total of 10 times, the stimulation intensity was 2mA, and the stimulation site was the cerebellum. The dosage of Xingnaojing was 20 ml each time by intravenous drip, diluted with 9% sodium chloride injection 200 ml, once a day. Intervention for two weeks.
  Interventions: Drug: XinNaoJing injection; Device: tDCS
- tDCS treatment group (Sham Comparator): The tDCS stimulation time was 20 minutes, once a day, 5 times a week, a total of 10 times, and the stimulation intensity was 2mA.
  Interventions: Device: tDCS
- XingNaoJing treatment group (Sham Comparator): The dosage of XingNaoJing was 20 ml each time by intravenous drip, diluted with 9% sodium chloride injection 200 ml, once a day.
  Interventions: Drug: XinNaoJing injection

INTERVENTIONS:
Drug: XinNaoJing injection — XingNaoJing injection is a kind of traditional Chinese medicine preparation, which has the effects of clearing heat and detoxifying, cooling blood and activating blood circulation, resuscitating the brain. In recent years, it has been often used in the treatment of related symptoms caused by qi and blood disturbance and cerebral blood stasis, and has achieved certain results. Xingnaojing injection contains Yujin to resuscitate phlegm, invigorate blood circulation and promote qi; Zhizi dissipates blood stasis and cleans heat; Both are subject medicine. Natural musk cleans the brain, Shujin Tongluo, Jun medicine; Borneol awaken awaken, for adjuvant. Small doses of musk restored brain function and improved cerebral circulation. Xingnaojing injection can promote the recovery of consciousness, reduce the level of plasma β-endorphin, and restore brain function. Borneol bi-dimensionally regulates the central nervous system, calms, prolongs the level of arousal, and protects the brain tissue.
  Arms: XingNaoJing treatment group; tDCS combined with XingNaoJing treatment group
Device: tDCS — tDCS stimulated the cerebellum for 20 minutes, once a day, 5 times a week, a total of 10 times, and the stimulation intensity was 2mA.
  Arms: tDCS combined with XingNaoJing treatment group; tDCS treatment group

SUMMARY:
The purpose of this study is to investigate the effect of tDCS stimulation of cerebellum combined with Xingnaojing on patients with disturbance of consciousness after craniocerebral injury, and to clarify the relationship between the following two points: (1) to clarify whether MMN, P300, fNIRS, BAEP, SEP can be used as objective indicators to distinguish VS from MCS. (2) To clarify the changes of consciousness level and brain function in DoC patients with craniocerebral injury treated with tDCS stimulation of cerebellum combined with Xingnaojing.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-80 years;
2. All patients met the diagnostic criteria of DoC;
3. more than 1 month after the initial head injury;
4. stable consciousness for at least 2 weeks before admission (no change in CRS-R total score);
5. no skull defect or large area of skull repair;
6. The legal representative authorized by the patient approved the experimental protocol and signed the informed consent form.

Exclusion Criteria:

1. supratentorial abnormalities on computed tomography (CT) or magnetic resonance imaging (MRI) involving more than one third of the middle cerebral artery territory;
2. a life expectancy of less than 3 months or a follow-up of less than 3 months;
3. retention of intracranial metal objects, cranial debridement, or presence of cranial defects and any clinically significant or unstable medical diseases;
4. EEG recording with significant muscle artifacts and inhibitory bursts;
5. nonconvulsive status epilepticus; Periodic or burst rhythms evoked by stimulation;
6. disturbance of consciousness due to surgical injury or tumor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
electroencephalogram | From enrollment to the end of treatment at 2 weeks
  Event-related potential: MMN and P300 in uV; Changes in power spectra and coherence and phase synchronization under delta, theta, and alpha in uV2.
Oxygenated hemoglobin concentration (HbO) | From enrollment to the end of treatment at 2 weeks
  Near-red function test fNRIS: to understand the changes of oxygen saturation in the head. HbO in uM.

SECONDARY OUTCOMES:
RLA grading Scale | From enrollment to the end of treatment at 2 weeks
  Purpose: Used to assess the level of consciousness in patients after brain injury, especially those in comatose or vegetative states.
  Scoring: The scale has 10 levels, each representing different levels of awareness and functioning.
  Level 1: No response (Coma) - No response to external stimuli. Level 2: Generalized response - Non-specific responses to stimuli. Level 3: Localized response - Specific responses to stimuli. Level 4: Confused-agitated - Disoriented and agitated behavior. Level 5: Confused-inappropriate - Inappropriate responses to commands, confusion.
  Level 6: Confused-appropriate - Appropriate responses but still confused. Level 7: Automatic-appropriate - Performs tasks automatically but still lacks flexibility.
  Level 8: Purposeful-appropriate - Independent with a certain level of awareness.
  Level 9: Purposeful-appropriate (standby assistance) - Increased independence. Level 10: Purposeful-appropriate (modified independent) - Fully independent.
Glasgow Coma Scale (GCS) | From enrollment to the end of treatment at 2 weeks
  Purpose: Assesses the neurological function and level of consciousness in patients, particularly those in a comatose state.
  Scoring: The scale evaluates three components: Eye response (E), Verbal response (V), and Motor response (M). Each component is scored from 1 to 4, and the total score is calculated.
  Eye response (E): 4 (spontaneous opening) to 1 (no response). Verbal response (V): 5 (oriented speech) to 1 (no response). Motor response (M): 6 (obeys commands) to 1 (no response). Total score: Ranges from 3 (deep coma) to 15 (fully alert and responsive).
Coma Recovery Scale-Revised (CRS-R) | From enrollment to the end of treatment at 2 weeks
  Purpose: Used to assess recovery in patients with severe brain injuries or in vegetative states.
  Scoring: Consists of 23 items evaluating different types of responses such as visual, auditory, and motor responses.
  Score range: 0 (no response) to 23 (full recovery). Components: The scale evaluates awareness, attention, perception, language, and motor responses.
FOUR Score (Full Outline of UnResponsiveness) | From enrollment to the end of treatment at 2 weeks
  Purpose: Used to assess the neurological status of patients with impaired consciousness, particularly those unable to communicate verbally.
  Scoring: Includes four parameters: Eye response, Brainstem reflexes, Respiratory pattern, and Motor response. Each parameter is scored from 0 to 4.
  Eye response: 0 (no response) to 4 (spontaneous eye opening). Brainstem reflexes: 0 (no reflexes) to 4 (normal reflexes). Respiratory pattern: 0 (no breathing) to 4 (spontaneous breathing). Motor response: 0 (no movement) to 4 (voluntary movement). Total score: Ranges from 0 (no response) to 16 (normal response).
Nutritional Risk Screening (NRS 2002) | From enrollment to the end of treatment at 2 weeks
  Purpose: Used to assess the nutritional risk of hospitalized patients. Scoring: The scale includes factors like disease severity, weight loss, and appetite.
  Disease severity: 0 (no disease) to 3 (severe disease). Appetite loss: 0 (no loss) to 3 (severe loss of appetite). Weight loss: 0 (no weight loss) to 3 (significant weight loss). Total score: A score of 3 or more indicates moderate to high nutritional risk.
Thrombosis Risk Assessment Scale (Padua Risk Assessment Scale) | From enrollment to the end of treatment at 2 weeks
  Purpose: Used to assess the risk of deep vein thrombosis (DVT) in hospitalized patients.
  Scoring: Includes clinical factors like age, obesity, cancer, and bed rest.
  Risk score: 0 (low risk) to 3 or more (high risk). Common factors: Advanced age, immobility, surgery, obesity, and malignancy are some factors that increase the risk.
Functional Independence Measure (FIM) | From enrollment to the end of treatment at 2 weeks
  Purpose: Assesses a patient's ability to perform activities of daily living, often used in rehabilitation settings.
  Scoring: Includes 13 items assessing daily living tasks (eating, dressing, bathing, toileting) and 5 cognitive tasks (social interaction, problem-solving).
  Score range: 1 (total dependence) to 7 (total independence). Total score: The lowest possible score is 18 (completely dependent) and the highest is 126 (completely independent).
Albumin | From enrollment to the end of treatment at 2 weeks
  Albumin in g/L
S100β | From enrollment to the end of treatment at 2 weeks
  S100β in ng/mL
NSE (Neuron-Specific Enolase) | From enrollment to the end of treatment at 2 weeks
  NSE (Neuron-Specific Enolase) in ng/mL
NFL (Neurofilament Light Chain) | From enrollment to the end of treatment at 2 weeks
  NFL (Neurofilament Light Chain) in pg/mL
Tau Protein | From enrollment to the end of treatment at 2 weeks
  Tau Protein in pg/mL
Ubiquitin Carboxy-terminal Hydrolase L1 (UCH-L1) | From enrollment to the end of treatment at 2 weeks
  Ubiquitin Carboxy-terminal Hydrolase L1 (UCH-L1) in ng/mL
GFAP (Glial Fibrillary Acidic Protein) | From enrollment to the end of treatment at 2 weeks
  GFAP (Glial Fibrillary Acidic Protein) in ng/mL
CK-MB (Creatine Kinase MB Isoform) | From enrollment to the end of treatment at 2 weeks
  CK-MB (Creatine Kinase MB Isoform) in U/L
ALT (Alanine Aminotransferase) | From enrollment to the end of treatment at 2 weeks
  ALT (Alanine Aminotransferase) in U/L
AST (Aspartate Aminotransferase) | From enrollment to the end of treatment at 2 weeks
  AST (Aspartate Aminotransferase) in U/L
Vitamin B12 | From enrollment to the end of treatment at 2 weeks
  Vitamin B12 in pg/mL
Thiamine (Vitamin B1) | From enrollment to the end of treatment at 2 weeks
  Thiamine (Vitamin B1) in nmol/L
Vitamin D | From enrollment to the end of treatment at 2 weeks
  Vitamin D in ng/mL
Phosphate | From enrollment to the end of treatment at 2 weeks
  Phosphate in mg/dL.

CONTACTS AND LOCATIONS:
Locations (1):
- Electroencephalography, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Yes